CLINICAL TRIAL: NCT04620772
Title: Efficacy and Safety of Cyclophosphamide in the Treatment of Refractory Proliferative Arachnoiditis in Central Nervous System Tuberculosis- A Randomized Double Blinded Placebo Controlled Trial
Brief Title: Cyclophosphamide in the Treatment of Refractory Proliferative Arachnoiditis in CNS Tuberculosis
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Arunmozhimaran Elavarasi, Dr Arunmozhimaran Elavarasi, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC-975/03.10.2020
Record Dates: First submitted 2020-10-27; First posted 2020-11-09 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Tuberculosis; Tubercular Meningitis; Arachnoiditis; Tuberculous (Etiology)
Keywords: tubercular optico-chiasmatic arachnoiditis; tubercular radiculo-myelitis
MeSH Terms: conditions — Tuberculosis; Tuberculosis, Meningeal; Arachnoiditis; Latent Tuberculosis | interventions — Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant, investigator, assessor and the statistician will be blinded to the treatment allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cyclophosphamide arm (Experimental): Participants randomized to the cyclophosphamide arm will be administered 750 mg/m2 body weight (rounded off to the nearest 50 mg above the calculated value) of cyclophosphamide diluted in normal saline every month (Total 6 months) along with equal dose of mesna 50% administered prior to infusion and 50% after the infusion of cyclophosphamide
  Interventions: Drug: Cyclophosphamide injection
- Placebo arm (Other): Participants randomized to the placebo group will be given similar quantity of normal saline and mesna as described above
  Interventions: Drug: Cyclophosphamide injection

INTERVENTIONS:
Drug: Cyclophosphamide injection — Cyclophosphamide vs placebo

SUMMARY:
Tubercular meningitis occurs in around 10% of those with extrapulmonary tuberculosis and is a major cause of mortality and morbidity. Inspite of effective Anti-tubercular drugs, still around 30% of patients develop complications due to arachnoiditis such as spinal tubercular radiculomyelitis, optico-chiasmatic arachnoiditis, development of new tuberculomas after starting therapy etc. which are probably immune mediated inflammatory responses due to paradoxical reaction to ATT.

The management of arachnoiditis is far from satisfactory. High dose methylprednisolone, intrathecal hyaluronic acid, thalidomide have been tried in small case series and case reports. However, the results have not been satisfactory.

There are two published reports of cyclophosphamide usage in TBM related vasculitis and stroke The investigators tried cyclophosphamide in four patients after consent, and found remarkable improvement in all of them. (Under peer review) In order to test this hypothesis, a randomized controlled trial is needed.

DETAILED DESCRIPTION:
Tubercular arachnoiditis occurring as a late complication of TBM is due to immune mediated reactions and is usually treated with high doses of corticosteroids. In the investigators' experience patients have received corticosteroids upto a duration of 20-28 months. In such cases, if the patient is refractory to corticosteroids, it is logical to step up to cyclophosphamide rather than continuing to give high dose steroids only similar to other immune mediated conditions such as CIDP, systemic and CNS vasulitis, Lupus nephritis etc.

Cyclophosphamide has been used most widely in the management of Lupus nephritis and maximum experience with the drug has been in this indication. So the dosage and duration of administration has been adapted from the induction phase dosing schedule of the ACR guidelines for the management of Lupus nephritis. The guidelines recommend 500 to 1000 mg/m2 BSA of cyclophosphamide. So the investigators decided to use 750 mg/m2 of the drug rounded off to the higher 50 mg.

Pathogenesis of tubercular arachnoiditis and Possible mechanism of cyclophosphamide Tubercular arachnoidiitis is a delayed complication in most cases due to inflammation in the optochiasmatic, spinal and other cranial nerves leading to neurologic deficits. In such situations, it is seen that there is an initial improvement in clinical symptoms followed by deterioration due to enlargement of lesions or appearance of new lesions, especially in patients with extrapulmonary tuberculosis. These new lesions are probably due to immune mediated mechanisms-it has been seen that in more than 95% of cases are drug sensitive and corticosteroids are the cornerstone of management of such patients. The complete pathogenesis of immune medicated tissue injury in tuberculosis has not been elucidated. Various studies have shown that there is an excess of pro-inflammatory cytokines and chemokines including TNF-alpha and interleukins that lead to recruitment of inflammatory cells and an exhuberant immune response in patients who develop these complications as compared to those who don't. There have been studies which have shown genetic polymorphisms in the genes encoding pro-inflammatory and anti-inflammatory cytokines-leading to difference in response to corticosteroids like LTA4 (Leukotriene- A4 hydrolase) gene. It is also well known that various immune mediated diseses such as SLE, multiple sclerosis etc are triggered by viruses and other infections. It is routine practice to treat acute bacterial meninigitis and tubercular meningitis with dexamethasone, which is again a steroid and immunosuppressant along with specific antibiotics or anti-tubercular therapy respectively based on evidence from systematic reviews and meta-analysis. Neurocysticercosis is treated with corticosteroids and other immunosuppressant medications such as methotrexate as recommended in guidelines, adalimumab and eternacept used as steroid sparing agents. Various other immune mediated complications of acute and chronic infections such as dengue myocarditis, ADEM etc are also treated with immunosuppression including corticosteroids. Lepra reactions in Leprosy are also treated using steroids, thalidomide, methotrexate, azathioprine, cyclophosphamide, cyclosporine etc.

In recent times, the corticosteroid- Dexamethasone has been shown to have mortality benefit in patients with moderate to severe COVID, proven in a randomized controlled trial. Simliarly, even though there are no RCT data, Tocilizumab, siltuximab and other immunosuppressant medications have been approved for emergency use based on their efficacy shown in large case series in COVID-19.

Justification for the use of cyclophosphamide this study:

Cyclophosphamide is a potent immunosuppressant agent. It is used in Lupus and other immune mediated conditions and has been shown to be effective in randomized controlled trials in Lupus nephritis, granulomatous polyangiiitis etc. Though it is widely used off label in various inflammatory immune mediated neurologic conditions such as CNS vasculitis, CIDP, multiple sclerosis, autoimmune encephalitis, refractory myasthenia gravis etc, the evidence for this is basically derived from the rheumatology and nephrology literature. It has to be emphasized that all the data for immunosuppression with azathioprine, cyclophosphamide, mycophenolate mofetil, methotrexate, calcineurin inhibitors in various immune mediated conditions have been derived from renal transplant/solid organ transplant cohorts, lupus nephritis cohorts, systemic vasculitis cohorts and inflammatory bowel disease cohorts. The various guidelines issued by the professional bodies for these conditions form the principles of treatment of rare conditions such as neuroimmunologic diseases. The major adverse effects of concern in patients on Cyclophosphamide is the occurrence of life threatening infections such as tuberculosis. It has been seen that patients on high dose corticosteroids and cyclophosphamide are at higher risk of infection than those on steroids alone or on neither drug.Though the risk of TB increases with administration of immunosuppressants, the mainstay of management is early diagnosis and starting appropriate therapy and not cessation of immunosuppression. In the context of SLE the occurrence of infection is also dependent on various other factors such as disease activity, previous exposure to tuberculosis etc. The Americal college of rheumatology guidelines do not say anything on the course of action in case patients develop infections. There are no professional guidelines for the management of infections in patients on cyclophosphamide. There are no RCTs on the most appropriate form of ATT regimens or the modification of immunosuppression in these conditions. There are various case series and case reports who have been systematically studied infections and their management including the large prospective EuroLupus cohort. None of these authors advice complete cessation of immunosuppression in patients who develop infections including tuberculosis. The guidelines for management of tuberculosis such as British thoracic society guidelines for the management of TB in CKD,do not suggest cessation of immunosuppression in post renal transplant patients. The guidelines clearly mention that TB in patients with CKD have to be treated in same lines of immunocompetent patients, and the anti-tubercular drugs may need to be given in renal modified doses. In case of tuberculosis risk, it has been shown by various long term follow up studies that a considerable proportion of patients with latent TB infections progress to develop active TB post transplantation or after treatment with immunosuppressants or biologic agents such as anti TNF therapy. In such circumstances, the guidelines suggest not dropping immunosuppression, but treatment of latent TB or active TB. The guidelines for the management of active TB in solid organ transplantation suggests early diagnosis and treatment of tuberculosis along with increasing the dose of immunosuppressants such as corticosteroids, cyclosporine or tacrolimus as the ATT regimen containing rifamycins tend to induce the metabolism of these immunosuppression and trough levels of calcineurin inhibitors have to be maintained by increasing the dose of cyclosporine or tacrolimus by upto 4-5 times.

These recommendations are mainly based on a large multicentre cohort of more than 2000 patients derived from 187 publications who had received solid organ transplantation and developed tuberculosis, where the dose of immunosuppressant drugs had been increased to maintain adequate blood levels to avoid rejection of the organ graft. Similar recommendations have been made by the TBNET consensus statement for management of Tuberculosis in transplant recipients.

The management of immunosuppression in these cases are mainly based on expert consensus in other conditions such as rheumatoid arthritis, spondyloarthropathy etc. The TBNET consensus statement also says that in case the organ is not vital or the infection is life threatening, it may be considered to reduce the level of immunosuppression. The guidelines for the use of anti TNF-α therapy is clearer in this aspect. While the occurrence of active TB during anti TNF-α therapy warrants withholding (NOT cessation) of immunosuppression, it may be re started 2 months after ATT the if patients demonstrate a favorable response to anti-TB therapy and require early resumption of anti TNF therapy.The BTS guidelines suggest that if active TB was diagnosed prior to starting of "Anti-TNF-α therapy, treatment should not be commenced for at least 2 months after antituberculosis treatment with full compliance has begun, supervised by a thoracic physician orinfectious disease specialist, and until the drug susceptibility profile of the organism in those with positive cultures is known, as a minimum." However, if the patient develops TB while on anti TNF therapy the anti-TNF-α treatment can be continued if clinically indicated because the patient would otherwise be prevented from receiving the continued clinical benefit to their underlying disease and may have a flare up or major clinical deterioration. The rationale provided by these guidelines is that HIV positive individuals with reduced CD4 counts and clinical TB, who are even more immunosuppressed than those on anti-TNF-a treatment, respond just as well to TB treatment as those who are HIV negative. Taking that logic forward, it may be reasonable to start therapy with cyclophosphamide three months after starting standard Anti tubercular therapy in patients with tubercular meningitis who have shown clearcut improvement followed by deterioration due to development of arachnoiditis and paradoxical immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending Neurology/Pulmonary Medicine/Medicine/Geriatric Medicine OPD/admitted in respective wards with proliferative tubercular arachnoiditis refractory to corticosteroids and standard Anti-tubercular drugs for CNS tuberculosis
* Atleast 14 years of age of all sexes
* Not more than 60 years of age at time of enrolment
* Patient was started on ATT for tubercular meningitis and had clearcut clinical improvement with resolution of fever/constitutional symptoms AND improvement in headache, vomiting and sensorium for atleast 10 days following which there is deterioration again due to arachnoiditis
* Developed paraparesis/quadriparesis/sphincter dysfunction due to spinal radiculomyelitis or vision loss due to due to optico-chiasmatic arachnoiditis with imaging evidence of arachnoiditis
* Has received standard ATT for atleast 3 months with adequate dose and compliance
* Received corticosteroids for treatment of arachnoiditis and deemed to be refractory to corticosteroids by the primary physician treating the patient
* MRI brain and spine are suggestive of Arachnoiditis
* CSF GeneXpert/Line Probe assay/cultures are not suggestive of drug resistant tuberculosis
* Reasonable clinical certainty OR allied investigations such as CECT chest/abdomen/PET CT ruling out drug resistant tuberculosis
* Other relevant investigations like CSF analysis not suggestive of alternative diagnosis such as cysticercal/ cryptococcal/other fungal infections/other causes of chronic meningitis such as brucella/ nocardia/ syphilis/recurrent viral meningitis/ carcinomatous/ lymphomatous meningitis or non infective causes such as sarcoidoisis/sub-arachnoid hemorrhage etc.
* Willing to undergo periodic assessment clinically and with MRI.
* Ready to provide consent for cyclophosphamide therapy
* Willing to adhere to protocol and comply with follow up visits

Exclusion Criteria:

* Not willing to provide consent
* Not willing to adhere to protocol
* Developed significant drug induced liver dysfunction so that patient is not being given Rifampicin, INH or pyrazinamide and is on modified ATT including quinolones, ethambutol and aminoglycosides or second line drugs only in the absence of Rifampicin and INH
* Drug resistant tubeculosis
* Men and Women of childbearing potential who are not using adequate contraception or women who are pregnant and lactating
* Patients who are on immunosuppressants such as cyclophosphamide/ azathioprine/ methotrexate/MMF/ calcineurin inhibitors for autoimmune conditions/post transplantation or chemotherapy for any systemic malignancy
* HBsAg, HIV serology and anti HCV positive
* Having life threatening infections such as pneumonia/urosepsis
* Patients who have developed large artery strokes with significant brain parenchymal damage
* Patients with expected life expectancy less than 1 year due to primary disease or comorbidity based on clinical prediction scores for specific disease
* Patients with systemic malignancy within the last 5 years
* Known allergy to cyclophosphamide or its preservatives/excipients
* Receiving cyclophosphamide for any indication in the last 12 weeks
* Gross hematuria prior to enrolment to the study/USG features of hemorrhagic cystitis
* Cytopenias Hct <25%, TLC<4000/mm3 or Platelet count <1,20,000/mm3 at the time of enrolment
* Alanine amino transferase (ALT) > 3 upper limit of normal at time of enrolment

Ages: 14 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional independece at 6 months | 6 months
  To compare the proportion of patients who attain functional independence (mRS-modified Rankin scale 0-2) 6 months after cyclophosphamide therapy for proliferative arachnoiditis refractory to corticosteroids and standard Anti-tubercular therapy in CNS tuberculosis to those who receive placebo.

SECONDARY OUTCOMES:
Independent ambulation | 6 months
  To compare the proportion of patients who attain independent ambulation 6 months after cyclophosphamide therapy for proliferative arachnoiditis refractory to corticosteroids and standard Anti-tubercular therapy in CNS tuberculosis to those who receive placebo.
Improvement in modified Rankin scale | 6 months
  To compare the proportion of patients improving from mRS ≥3 to mRS ≤2 six months post cyclophosphamide therapy
Improvement in visual acuity (1) | 6 months
  To compare the proportion of patients who attain atleast 2 points improvement on Snellen's chart in visual acuity 6 months after cyclophosphamide therapy for proliferative arachnoiditis refractory to corticosteroids and standard Anti-tubercular therapy in CNS tuberculosis to those who receive placebo.
Improvement in visual acuity (2) | 6 months
  To compare proportion of patients who attain atleast two point improvement on a semiquantitative visual acuity measurement in those who have visual acuity less than 1/60 on snellen's chart (finger counting at 1 m, hand movements at 1 m, perception of light, no perception of light considered as discrete points below 1/60 vision on standard Snellen's chart) 6 months after cyclophosphamide therapy
Improvement in visual acuity (3) | 6 months
  To compare proportion of patients improving from visual acuity of <3/60 in the better eye to 3/60 or more 6 months post cyclophosphamide therapy
Improvement in sphincter function | 6 months
  To compare the proportion of patients who attain improvement in bladder/bowel function 6 months after cyclophosphamide therapy for proliferative arachnoiditis refractory to corticosteroids and standard Anti-tubercular therapy in CNS tuberculosis to those who receive placebo..
Change in mRS | 6 months
  Shift analysis pre-and 6 months post therapy in terms of change in mRS
Patient well being | 6 months
  Comparing Global patient well being as assessed by SF-36 pre and 6 months post cyclophosphamide therapy
Life threatening infections | 3 months
  Occurrence of life threatening infections necessitating cessation of therapy upto 3 months post cyclophosphamide therapy
Infections needing hospitalization | 3 months
  Occurrence of infections needing hospitalization or intravenous antibiotic/antiviral/anti-fungal therapy upto 3 months post cyclophosphamide therapy
Flare up of TB | 3 months
  Flare up of underlying tuberculosis upto 3 months post cyclophosphamide therapy
Cytopenias | 6 weeks
  Occurrence of Grade III cytopenias defined as per common terminology criteria for adverse events v 5.0 upto 6 weeks post cyclophosphamide therapy
Transaminitis | 6 weeks
  Grade III transaminitis as per CTCAE v 5.0 upto 6 weeks post cyclophosphamide therapy
Hemorrhagic cystitis | 2 weeks
  Occurrence of hemorrhagic cystitis upto 2 weeks post cyclophosphamide therapy
Adverse effects | 3 months
  Any other significant adverse effect

IPD SHARING:
Plan to Share IPD: Undecided
Based on Institutional protocol

REFERENCES:
- [Background] Goyal V, Elavarasi A, Abhishek, Shukla G, Behari M. Practice Trends in Treating Central Nervous System Tuberculosis and Outcomes at a Tertiary Care Hospital: A Cohort Study of 244 Cases. Ann Indian Acad Neurol. 2019 Jan-Mar;22(1):37-46. doi: 10.4103/aian.AIAN_70_18. PMID 30692758
- [Background] Gonzalez-Duarte A, Higuera-Calleja J, Flores F, Davila-Maldonado L, Cantu-Brito C. Cyclophosphamide treatment for unrelenting CNS vasculitis secondary to tuberculous meningitis. Neurology. 2012 Apr 17;78(16):1277-8. doi: 10.1212/WNL.0b013e318250d84a. Epub 2012 Apr 4. No abstract available. PMID 22491870
- [Background] Celotti A, Vianello F, Sattin A, Malipiero G, Faggin R, Cattelan A. Cyclophosphamide immunomodulation of TB-associated cerebral vasculitis. Infect Dis (Lond). 2018 Oct;50(10):779-782. doi: 10.1080/23744235.2018.1467038. Epub 2018 Apr 28. No abstract available. PMID 29708006